CLINICAL TRIAL: NCT01966757
Title: Neuronal Ceroid Lipofuscinosis and Associated Sleep Abnormalities
Status: Completed | Type: Observational
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Lenora Lehwald, Assistant Professor of Clinical Pediatrics, Nationwide Children's Hospital
Other Study IDs: IRB13-00376
Record Dates: First submitted 2013-09-25; First posted 2013-10-22 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Neuronal Ceroid Lipofuscinosis; Batten's Disease
Keywords: Neuronal Ceroid Lipofuscinosis; NCL; Batten's Disease; Children's Sleep Habits Questionnaire; Restless Leg Syndrome
MeSH Terms: conditions — Neuronal Ceroid-Lipofuscinoses; Restless Legs Syndrome

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Neuronal ceroid lipofuscinosis patients: Caregiver of patient with NCL to provide information regarding patient's sleep habits

SUMMARY:
Neuronal Ceroid Lipofuscinosis (NCL) also known at Batten's disease is the most common neurodegenerative disorder in children. Families often report the patient has a sleep disturbance. This is a questionnaire to be completed by the family to better understand the sleep pattern and sleep difficulties experienced by individuals who have been diagnosed with NCL.

DETAILED DESCRIPTION:
Neuronal Ceroid Lipofuscinosis (NCL) is the most common neurodegenerative disorder in children characterized by seizures, blindness, ataxia, myoclonia and loss of cognition. There are 12 clinical types identified with a concurrent genetic abnormality. The diagnosis is determined by gene testing and skin biopsy findings although genetic testing has supplanted skin biopsy in most cases. Numberous studies have confirmed the presence of sleep disorder in patients with NCL but these cases were documented over a decade ago. The investigators would like to study the prevalence of sleep disorders in this group of patients. The investigators will distribute a Children's Sleep Habits Questionnaire (CSHQ) to the family of the patient to complete and provide a information regarding the patient's sleep. In addition to the validated sleep questionnaire a separate demographic questionnaire will be given to the family to identify the type of NCL, presence or absence of blindness, presence or absence of seizures, interventions tried to treat sleep disturbance. The last questions of the study are asking for the presence or absence of Restless Leg Syndrome symptoms.

ELIGIBILITY:
Inclusion Criteria:

* patient with a known diagnosis of Neuronal Ceroid Lipofuscinosis (NCL) by DNA or electron microscopy studies Family member completing study must be able to read and understand the Children's Sleep Habits Questionnaire (CSHQ) and Demographic questions

Exclusion Criteria:

* patient without a confirmed diagnosis of NCL Family member completing the study is unable to read and understand the questionnaires

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with a known diagnosis of Neuronal Ceroid Lipofuscinosis by biopsy or genetic testing
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2013-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Sleep disturbance | one year
  Identify the presence of sleep disturbance in children with Neuronal Ceroid Lipofuscinosis using the Children's Sleep Habits Questionnaire (CSHQ) and using the 8 subscales further identify specific areas of difficulty

SECONDARY OUTCOMES:
Epilepsy onset | one year
  Correlate the onset of sleep difficulties with history of epilepsy
Blindness | one year
  Correlate the onset of sleep difficulties with loss of vision

CONTACTS AND LOCATIONS:
Overall Officials: Lenora M Lehwald, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Owens JA, Spirito A, McGuinn M. The Children's Sleep Habits Questionnaire (CSHQ): psychometric properties of a survey instrument for school-aged children. Sleep. 2000 Dec 15;23(8):1043-51. PMID 11145319
- [Result] Lehwald LM, Pappa R, Steward S, de Los Reyes E. Neuronal Ceroid Lipofuscinosis and Associated Sleep Abnormalities. Pediatr Neurol. 2016 Jun;59:30-5. doi: 10.1016/j.pediatrneurol.2016.02.009. Epub 2016 Mar 3. PMID 27105763